CLINICAL TRIAL: NCT03644108
Title: A Phase I, Open-label, Single-dose, Single-Period Study to Evaluate the Pharmacokinetics of Mucinex® 600 mg Extended-Release Bi-layer Tablet in Normal Healthy Subjects.
Brief Title: Study to Evaluate the Pharmacokinetics of Mucinex 600 mg Extended-release Bi-layer Tablet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser Inc. (Industry)
Responsible Party: Sponsor
Organization: Reckitt Benckiser LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-GGE-04
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Guaifenesin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mucinex® ER 600 mg (Experimental): Single dose of Mucinex® 600 mg Extended-Release (ER) Bi-Layer tablet taken with 240 mL of water after an overnight fast
  Interventions: Drug: Mucinex® ER 600 mg

INTERVENTIONS:
Drug: Mucinex® ER 600 mg — Single dose of Mucinex® 600 mg ER Bi-Layer tablet
  Other Names: guaifenesin

SUMMARY:
Evaluate the Pharmacokinetics of Mucinex® 600 mg Extended-Release Bi-Layer Tablet in Normal Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females between the ages of 19 and 55 years, inclusive.
2. Females of childbearing potential must have been using 1 of the following acceptable birth control methods:

   1. Intra-uterine device (IUD) in place for at least 3 months prior to Day 1 through 30 days beyond study completion or first menstrual period.
   2. Barrier method (condom or diaphragm) with spermicide for at least 7 days prior to screening through 30 days beyond study completion or first menstrual period (whichever is longer).
   3. Stable hormonal contraceptive (e.g., PO, depo injection, transdermal patch, or vaginal ring) for at least 3 months prior to Day 1 through 30 days beyond completion of study or first menstrual period.

   Note: Abstinence is not an acceptable form of contraception; however, abstinent female subjects may have been admitted to the study if they agreed, and signed a statement to the effect, that upon becoming sexually active, would use a condom with spermicide from screening through 30 days beyond completion of the study.
3. Females of non-childbearing potential must have been surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to Day 1 or hysterectomy and/or bilateral oophorectomy at least 3 months prior to Day 1) or postmenopausal >2 years prior to Day 1. A follicle stimulating hormone (FSH) level >40 miU/mL must be obtained and recorded for any postmenopausal females.
4. Good general health as determined by the PI's review of medical history, physical examination, vital sign measurements, electrocardiogram (ECG), and clinical laboratory measures.
5. Within 15% of ideal body weight (Table of 'Desirable Weights of Adults' Metropolitan Life Insurance Company, 1983).
6. Non-tobacco users, who had not used nicotine or nicotine-containing products for at least 365 days prior to Day 1.
7. Able to read, understand, and sign the informed consent form (ICF), after the nature of the study had been explained.
8. Negative urine screen for drugs of abuse and alcohol at screening and each check-in.
9. If female, negative finding on serum pregnancy test at screening and each check-in.

Exclusion Criteria:

1. Clinically significant abnormalities detected by medical history, physical examination, vital sign measurements, ECG, or clinical laboratory findings (as determined by the PI/designee) including a hemoglobin value <12 g/dL at screening. If a subject's hemoglobin drops below 11.0 g/dL during the study, the subject may be dropped from the study at the discretion of the PI.
2. Any disease or condition that could impact absorption, distribution, metabolism, or elimination of the study drugs (as determined by the PI/designee).
3. Alcoholism or medicinal product or drug abuse within the past 2 years or excessive alcohol consumption (more than 10 units per week) (1 unit is defined as 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of spirits (i.e., 'hard' liquor such as gin, whiskey, or vodka, et. al.). The subject could not experience tolerance, withdrawal, compulsive use, or substance related problems such as medical complications, disruption in social and family relationships, vocational or financial difficulties, or legal problems.
4. Females who were pregnant or nursing.
5. History of hypersensitivity reaction to guaifenesin.
6. Receipt of an investigational drug within 30 days prior to Day 1.
7. Abnormal diet (for whatever reason) during the 30 days prior to Day 1.
8. Donation of blood or significant loss of blood within 56 days or plasma within 14 days prior to Day 1.
9. Known or suspected use of illicit drugs.
10. The use of any medication (with the exception of hormonal contraceptives for women of childbearing potential) for 14 days or 5 half-lives of the drug (whichever is longer) prior to Day 1.
11. Test positive for Hepatitis B surface antigen, Hepatitis C antibodies, or human immunodeficiency virus (HIV).

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06-04 (Actual); Primary Completion 2009-06-15 (Actual); Study Completion 2009-06-15 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-centre study.
Pre-assignment Details: A total of 30 subjects were screened for the study; All 30 subjects were included single-period.
Groups:
- Mucinex® 600 mg ER: Single dose Mucinex® 600 mg Extended-Release (ER) Bi-Layer tablet expectorant by mouth.
Period: Overall Study
Arm/Group | Mucinex® 600 mg ER
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mucinex® 600 mg ER
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race [Count of Participants; unit: Participants]
  Asian | 1
  Black | 2
  Caucasian | 27
Weight [Mean (Standard Deviation); unit: lb] | 160.4 (23.11)
Height [Mean (Standard Deviation); unit: in] | 68.41 (3.222)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.976 (1.8368)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Guaifenesin
Description: Pharmacokinetic Parameters Cmax (Maximum observed drug concentration)
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14, 16 and 24 hours (post-dose) on Day 1 and 2
Population: Data Sets Analyzed as all 30 subjects were included in the guaifenesin concentration tables and the calculation of guaifenesin Pharmacokinetic (PK) parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mucinex® 600 mg ER
Number analyzed (Participants) | 30
ng/mL | 876 (45.1)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUC(0-t)) of Guaifenesin
Description: Area under the drug concentration-time curve calculated using linear trapezoidal summation from time zero to time t, where t is the time of the last measurable concentration (Ct).
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng∙hr/mL
Arm/Group | Mucinex® 600 mg ER
Number analyzed (Participants) | 30
ng∙hr/mL | 3670 (45.4)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC(0-inf)) of Guaifenesin
Description: Area under the drug concentration-time curve from time zero to infinity, AUC(0-inf) = AUC(0-t) + Ct/Kel, where Kel is the terminal elimination rate constant.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng∙hr/mL
Arm/Group | Mucinex® 600 mg ER
Number analyzed (Participants) | 30
ng∙hr/mL | 3694 (45.2)

4. Primary Outcome: Time to Maximum Observed Concentration (Tmax) of Guaifenesin
Description: Pharmacokinetic Parameter tmax (Time of the maximum observed drug concentration).
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Mucinex® 600 mg ER
Number analyzed (Participants) | 30
hr | 0.752 [0.498 to 2.00]

5. Primary Outcome: Area Under Plasma Concentration Curve Ratio (AUCR) of Guaifenesin
Description: Ratio of AUC(0-t) to AUC(0-inf), referred to as AUCR. [AUCR = AUC(0-t) / AUC(0-inf)]
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mucinex® 600 mg ER
Number analyzed (Participants) | 30
Ratio | 0.9934 (0.007125)

6. Primary Outcome: Apparent Terminal Elimination Rate Constant (Kel) of Guaifenesin
Description: Apparent terminal elimination rate constant (Kel) calculated by linear regression of the terminal linear portion of the log concentration-time curve.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Mucinex® 600 mg ER
Number analyzed (Participants) | 30
1/hr | 0.455 (0.200)

7. Primary Outcome: Apparent Terminal Elimination Half-life (t1/2) of Guaifenesin
Description: Apparent terminal elimination half-life (t1/2) calculated as ln(2)/Kel.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Mucinex® 600 mg ER
Number analyzed (Participants) | 30
hr | 1.91 (1.11)

8. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: Intensity was determined by the Investigator. For symptomatic AEs the following definitions were applied.
  Mild = AE did not limit usual activities; subject may have experienced slight discomfort.
  Moderate = AE resulted in some limitation of usual activities; subject may have experienced significant discomfort.
  Severe = AE resulted in an inability to carry out usual activities; subject may have experienced intolerable discomfort/pain.
  Relationship to Investigational Medicinal Products (IMP)
  Unlikely = Slight, but remote, chance that AE was caused by IMP. Possible = Reasonable suspicion that the AE was caused by IMP. Probable = Most likely that AE was caused by IMP.
Time Frame: Up to Day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mucinex® 600 mg ER
Number analyzed (Participants) | 30
Participants
  TEAE by severity: Mild | 5
  TEAE by severity: Moderate | 0
  TEAE by severity: Severe | 0
  Relationship to IMP - Unlikely | 5
  Relationship to IMP - Possible | 0
  Relationship to IMP - Probable | 0

ADVERSE EVENTS:
Time Frame: Up to Day 2
Arm/Group | Mucinex® 600 mg ER
All-Cause Mortality (participants affected / at risk) | 5/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 5/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mucinex® 600 mg ER (N=30)
Headache (Nervous system disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No